CLINICAL TRIAL: NCT03789942
Title: Comparative Clinical Study of Cardiac and Respiratory Modifications Produced in Patients Undergoing Oral Surgery Through Local Anesthesia, Local Anesthesia and Oral Sedation With Midazolam, and Local Anesthesia Associated to Nitrous Oxide.
Brief Title: Modification of Blood Pressure Levels and Oxygen Saturation in Patients Undergoing Conscious Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Luis Ortiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ÉTICA-ULE-011-2016
Record Dates: First submitted 2018-07-14; First posted 2018-12-31 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2018-12

CONDITIONS: Dental Anxiety
MeSH Terms: interventions — Surgery, Oral

STUDY DESIGN:
Intervention Model Description: 90 patients will be randomly divided into three groups of 30 patients each. They will be given a prior consent both of the procedures to be performed and of the sedation procedure to which they will be subjected, if that is the case, without knowing what dose they will be administered. In case of being sedated, they will be informed verbally of the details concerning the procedure.
  Group 1, 30 patients treated by Oral Surgery procedures exclusively with Local Anesthesia.
  Group 2, 30 patients treated by procedures of Oral Surgery with Local Anesthesia and Oral Sedation with Midazolam.
  Group 3, 30 patients treated by Oral Surgery procedures with Local Anesthesia and Inhalation Sedation with a mixture of Nitrous Oxide / Oxygen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1. Local anaesthesia for oral surgery (Active Comparator): Administration of local anesthesia, 40mg.epinephrine once. Oral surgery procedures Suturing End of procedure
  Interventions: Procedure: Oral surgery
- 2. Local anesthesia with Midazolam (Active Comparator): Administration of 40mg. epinephrine once, and Oral Sedation with Midazolam 0,5 mgr per kilo once.
  Oral surgery procedures Suturing End of procedure
  Interventions: Procedure: Oral surgery
- 3. Local anesthesia and sedation (Active Comparator): Administration of 40mg. epinephrine once, and Inhalation Sedation by Nitrous Oxide / Oxygen.
  Nitrous oxide sedation Oral surgery procedures Suturing End of procedure Reduce nitrous oxide concentration
  Interventions: Procedure: Oral surgery

INTERVENTIONS:
Procedure: Oral surgery — Oral surgery procedures

SUMMARY:
The objective is to compare the changes produced in cardiological and respiratory parameters in three groups of patients undergoing oral surgery. The first group was treated with local anesthesia, a second group with local anesthesia plus oral conscious sedation with midazolam, and a third subject under anesthesia local with inhalation sedation with nitrous oxide.

A total of 90 non-cooperative phobic adult patients belonging to the group of patients of the University Master in Oral Surgery, Implantology and Periodontics of the University of León will be included in this study, after their information and acceptance of verbal and written consent, separated into three groups without significant differences in age, sex, smoking habits, cardiac or respiratory pathologies, and will be treated by advanced procedures of Oral Surgery, Periodontics and Implantology such as Sinus lift, Periodontal Surgeries and Implant Surgeries.

They will be randomly divided into three groups of 30 patients each. They will be given a prior consent both of the procedures to be performed and of the sedation procedure to which they will be subjected, if that is the case, without knowing what dose they will be administered. In case of being sedated, they will be informed verbally of the details concerning the procedure.

DETAILED DESCRIPTION:
A total of 90 non-cooperative phobic adult patients will be included in this study, after their information and acceptance of verbal and written consent, separated into three groups without significant differences in age, sex, smoking habits, cardiac or respiratory pathologies, and will be treated by advanced procedures of Oral Surgery, Periodontics and Implantology such as Sinus lift, Periodontal Surgeries and Implant Surgeries.

Initially, a complete health questionnaire will be filled out in all patients, and Partial Oxygen Saturation (SpO2), Respiratory Rate, Respiratory Volume in the form of Forced Vital Capacity (FVC), and also Forced Expiration Volume will be recorded as respiratory records (FEV) and Maximum Expiratory Flow (PEF), and as cardiac registers the Heart Rate, and the Systolic and Diastolic Blood Pressure before starting the procedure, records that will be repeated every 5 minutes during and until the end of it. The parameters will be recorded every 5 minutes, except for the parameters VFC, FEV1 and PEF that will be recorded exclusively at the beginning and at the end of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of phobic patients
* Not having contraindications to be anesthetized or sedated, and
* Present an acceptable state of health (ASA I and ASA II).

Exclusion Criteria:

* Clinical conditions; ASA III, ASA IV and ASA V

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Partial Oxygen Saturation (SpO2) change | From the beginning of the sedation until the end, assessed Up to one hour
  Partial Oxygen Saturation (SpO2) change
Respiratory Rate change | From the beginning of the sedation until the end, assessed Up to one hour
  Respiratory Rate change
Forced Vital Capacity (FVC) change | From the beginning of the sedation until the end, assessed Up to one hour
  Forced Vital Capacity (FVC) change
Forced Expiration Volume (FEV) change | From the beginning of the sedation until the end, assessed Up to one hour
  Forced Expiration Volume (FEV) change
Maximum Expiratory Flow (PEF) change | From the beginning of the sedation until the end, assessed Up to one hour
  Maximum Expiratory Flow (PEF) change
Heart Rate change | From the beginning of the sedation until the end, assessed Up to one hour
  Heart Rate change
Diastolic Blood Pressure change | From the beginning of the sedation until the end, assessed Up to one hour
  Diastolic Blood Pressure change
Systolic blood pressure change | From the beginning of the sedation until the end, assessed Up to one hour
  Systolic blood pressure change

CONTACTS AND LOCATIONS:
Overall Officials: ORTIZ CAMARERO, Principal Investigator — ASISTANT PROFESSOR
Locations (1):
- Clinica Luis Ortiz, Burgos, Spain